CLINICAL TRIAL: NCT04784065
Title: A Pilot Randomized Controlled Trial for Hand Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Grace Hsiao-Wei Lo, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H44508
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Hand Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The occupational therapists fabricating the orthoses used the study are the only ones not blinded in this study. The participants, principal investigator, and research assistants are all blinded to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment arm with control orthosis (Active Comparator): A resting orthosis that was modified to allow for convenient application of finger traps. A finger trap was customized to the most symptomatic DIP and any other digit that the participant requested.
  The participants were asked to continue the orthosis schedule for the full 24 weeks of the study. Besides the resting hand orthosis, the SOC treatment included a thermal modality, activity modification/ joint protection education, and range of motion exercises.
  Interventions: Device: Hand orthosis
- Treatment arm with experimental orthosis (Experimental): An identical resting hand orthosis to what the traction arm received without the finger trap modifications.
  The participants were asked to continue the orthosis schedule for the full 24 weeks of the study. Besides the resting hand orthosis, the SOC treatment included a thermal modality, activity modification/ joint protection education, and range of motion exercises.
  Interventions: Device: Hand orthosis

INTERVENTIONS:
Device: Hand orthosis — An orthosis applied to a hand affected by osteoarthritis with the expectation that it will improve symptoms and possibly structural progression.

SUMMARY:
This is a study involving people receiving care at the Michael E. DeBakey VA Medical Center, Houston Texas. We are studying people who have hand osteoarthritis (the most common form of arthritis that involves the hand) and testing treatments for the condition with the hope that we can help to improve hand pain as well as limit the damage that occurs related to the arthritis. People who choose to participate, are randomly assigned to one of two treatments, both expected to be helpful.

DETAILED DESCRIPTION:
The research will be conducted at the following location(s):

Baylor College of Medicine, Baylor St. Luke's Medical Center (BSLMC), and Michael E. DeBakey Veterans Affairs Medical Center.

Participants of this study are consented for the study, randomized into one of two treatment groups for hand osteoarthritis, both expected to improve hand symptoms. At the beginning of the study, many questionnaires, a physical exam, photographs of the hands, some x-rays, on a limited few people, and MRI will be obtained. Then the participants will be provided treatments for hand osteoarthritis based on the group wo which they were randomly assigned. One aspect of one of the treatments is viewed as experimental but the risks related to the treatment are considered to be low, so the risk-benefit ratio for participation in this study are good. We see patients in follow up more frequently during the first month, and then at 3 months and then 6 months of follow up. At the final visit, we will repeat the xrays and the MRIs.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled to receive medical care at the Michael E. DeBakey VA Medical Center
* At least 3 joints affected by distal interphalangeal (DIP) nodal hand OA
* DIP nodal hand OA will be defined as Heberden's nodes on physical exam.
* Sufficiently severe frequent pain of at least one DIP
* Frequent pain: pain on most days of the month for at least one month in the last year.
* Minimum VAS pain severity of 40 on a 0 - 100 scale

Exclusion Criteria:

* History or current inflammatory arthritides (examples: gout, psoriatic arthritis, and rheumatoid arthritis)
* Prior surgery on the DIP joints
* Planned surgery for the DIP joints
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace H Lo, MD MSc, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - NYU Langone, New York, New York
  - Michael E. DeBakey VA Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data from this study may be requested from other researchers 3 years after the completion of the primary endpoint by contacting Dr. Grace Lo.
Supporting Information: ICF
Time Frame: 3 years after the completion of the primary endpoint
Access Criteria: To be determined on a case by case basis.

REFERENCES:
- See also: Presented at the American College of Rheumatology Convergence Meeting, Nov 2024. — https://acrabstracts.org/abstract/a-pilot-randomized-controlled-trial-for-hand-osteoarthritis/

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm With Control Orthosis: Identical resting hand orthosis to what the traction arm received without the finger trap modifications.
  The participants were asked to continue the orthosis schedule for the full 24 weeks of the study. Besides the resting hand orthosis, the SOC treatment included a thermal modality, activity modification/ joint protection education, and range of motion exercises.
- Treatment Arm With Experimental Orthosis: A resting orthosis that was modified to allow for convenient application of finger traps. A finger trap was customized to the most symptomatic DIP and any other digit that the participant requested.
  The participants were asked to continue the orthosis schedule for the full 24 weeks of the study. Besides the resting hand orthosis, the SOC treatment included a thermal modality, activity modification/ joint protection education, and range of motion exercises.
Period: Overall Study
Arm/Group | Treatment Arm With Control Orthosis | Treatment Arm With Experimental Orthosis
Started | 17 | 16
Completed | 8 | 13
Not Completed | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm With Control Orthosis | Treatment Arm With Experimental Orthosis | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.5 (7.1) | 65.2 (6.6) | 65.8 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 7 | 10 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 10 | 17
  White | 9 | 5 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Study Hand VAS [Mean (Standard Deviation); unit: Units on a scale] | 69.3 (18.9) | 59.4 (20.0) | 64.5 (19.8)

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) for Pain in the More Symptomatic Hand That Includes the Most Symptomatic DIP Joint by 24 Weeks of Use of Traction Therapy With Standard of Care Treatment for Hand OA to Establish Efficacy of Traction Therapy.
Description: An assessment of pain intensity in a given hand. - high values are worse outcomes.
  Minimum score = 0 Maximum score = 100
Time Frame: 24 week follow up
Population: All randomized participants
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Arm With Control Orthosis | Treatment Arm With Experimental Orthosis
Number analyzed (Participants) | 17 | 16
units on a scale | -16.1 [-31.3 to -0.8] | -15.7 [-30.0 to -1.4]

2. Primary Outcome: The Primary Structure Endpoint Will be Change in Sum of the Kellgren and Lawrence Score of All Distal InterPhalangeal Joints in the Hand That Was Placed in an Orthosis Over 24 Weeks.
Description: An assessment of radiographic OA severity. (high values are worse outcomes) Minimum score = 0 Maximum score = 16
Time Frame: 24 week follow up
Population: Those participants at the Houston site who were randomized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Arm With Control Orthosis | Treatment Arm With Experimental Orthosis
Number analyzed (Participants) | 11 | 12
units on a scale | 0 (0) | 0 (0)

3. Secondary Outcome: The Functional Index for Hand Osteoarthritis (FIHOA)
Description: An assessment of hand function. (high values are worse outcomes) Minumum score = 0 Maximum score = 30
Time Frame: 24 week follow up
Population: All those randomized.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Arm With Control Orthosis | Treatment Arm With Experimental Orthosis
Number analyzed (Participants) | 17 | 16
units on a scale | 0.6 [-2.9 to 4.2] | -2.6 [-5.1 to -0.2]

4. Secondary Outcome: The Disabilities of Arm Shoulder and Hand (DASH)
Description: An assessment of hand disability. (high values are worse outcomes) Minimum score = 30 Maximum score = 150
Time Frame: 24 week follow up
Population: All those randomized.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Arm With Control Orthosis | Treatment Arm With Experimental Orthosis
Number analyzed (Participants) | 17 | 16
units on a scale | 0.9 [-6.9 to 8.7] | -9.9 [-17.9 to -2.0]

5. Secondary Outcome: Functional Dexterity Test
Description: An assessment of hand functional dexterity. (high values are worse outcomes) Measure of the number of seconds it takes for the participant to complete a series of activities. Penalty scores are assigned if the quality of the activity performed is imperfect.
  Minimum score = 0 Maximum score = indefinite
Time Frame: 24 week follow up
Population: All participants who were randomized.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Treatment Arm With Control Orthosis | Treatment Arm With Experimental Orthosis
Number analyzed (Participants) | 17 | 16
seconds | -3.8 [-11.8 to 4.3] | -6.4 [-11.0 to -1.9]

6. Secondary Outcome: Grip Strength
Description: An assessment of the amount of force that can be applied with grip. (low values are worse outcomes)
Time Frame: 24 week follow up
Population: All randomized.
Measure: Mean (95% Confidence Interval); unit: pounds
Arm/Group | Treatment Arm With Control Orthosis | Treatment Arm With Experimental Orthosis
Number analyzed (Participants) | 17 | 16
pounds | 3.1 [-0.5 to 6.7] | 5.3 [1.5 to 9.1]

7. Secondary Outcome: Pinch Strength
Description: An assessment of the amount of force that can be applied with pinching between thumb and the 2nd and 3rd fingers. (low values are worse outcomes)
Time Frame: 24 week follow up
Population: All randomized.
Measure: Mean (95% Confidence Interval); unit: pounds
Arm/Group | Treatment Arm With Control Orthosis | Treatment Arm With Experimental Orthosis
Number analyzed (Participants) | 17 | 16
pounds | 0.4 [-1.3 to 2.0] | 0.2 [-0.8 to 1.3]

8. Secondary Outcome: The Number of DIP Joints That Exhibit Tenderness in the Study Hand
Description: The number of DIP joints that exhibit tenderness (dichotomously assessed - yes/no) in the study hand. (high values are worse outcomes) Minimum score = 0 Maximum score = 4
Time Frame: 24 week follow up
Population: All randomized
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment Arm With Control Orthosis | Treatment Arm With Experimental Orthosis
Number analyzed (Participants) | 17 | 16
score on a scale | -0.2 [-0.7 to 0.4] | -0.4 [-1.1 to 0.2]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment Arm With Control Orthosis | Treatment Arm With Experimental Orthosis
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 8/17 | 8/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm With Control Orthosis (N=17) | Treatment Arm With Experimental Orthosis (N=16)
Discomfort from the orthosis (Musculoskeletal and connective tissue disorders) | 5 (9) | 7 (9)
Skin Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin blistering (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Numbness/Tingling (Nervous system disorders) | 5 (6) | 1 (1)
Fall (Nervous system disorders) | 0 (0) | 1 (1)
Elective surgery to repair incisional hernia (Eye disorders) | 0 (0) | 1 (1)
Thoracic spine pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Knee injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT04784065/Prot_SAP_000.pdf